CLINICAL TRIAL: NCT05262036
Title: The Effects of a Longevity Supplement on Skin Health, Blood Biomarkers and Mental Health
Brief Title: The Effects of a Longevity Supplement on Aging and Photoaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: AgeLess Sciences Inc. (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Integrative Dermatologist, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NS-1
Record Dates: First submitted 2022-02-13; First posted 2022-03-02 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Photoaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-aging Supplement (Experimental): Mixture (powder) of vitamins and nutrients
  Interventions: Dietary Supplement: Anti-aging Supplement
- Placebo excipients (Placebo Comparator): All excipients in powder WITHOUT vitamins and nutrients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anti-aging Supplement — Mixture of different vitamins and nutrients
  Arms: Anti-aging Supplement
Dietary Supplement: Placebo — Excipient powder
  Arms: Placebo excipients

SUMMARY:
This study evaluates the use of an oral supplement to see if it can shift the function of the skin and the appearance of fine lines and wrinkles, its impact on biomarkers associated with aging, and its impact on mental health.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects
* Subjects who are between the ages of 35 to 70.
* Subjects must be able to read and comprehend study procedure and consent forms
* Must be willing to comply with all protocol requirements
* Must be willing to have facial photographic images taken

Exclusion Criteria:

* Women who have been pregnant in the last three months, currently pregnant, preparing to become pregnant during the study, or breastfeeding.
* Individuals who have a history of smoking or chewing tobacco or vaping nicotine based product within the past year or if the pack-year history of smoking tobacco is greater than 5 pack-years.
* Those that have undergone a change in hormone-based therapies such as, but not limited to, oral contraceptive pills or progesterone pills within the last 2 months. Progesterone releasing IUDs are considered hormone-based therapy. Spironolactone is not considered a hormone-based therapy.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.
* Subjects who have a history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study in the opinion of the principal investigator.
* Has a skin disease on the face that will interfere with image collection and assessment in the opinion of the investigator.
* History of any significant chronic disease including endocrine, inflammatory, cardiovascular, renal, liver, gastro-intestinal, psychiatric, neurological, neoplastic, or metabolic disease for at least 90 days prior to screening. Clinical significance of active disease will be assessed by the Qualified Investigator to determine eligibility.
* Subjects with or who have recently experienced traumatic injury, infections, or major surgery at the discretion of the Qualified Investigator.
* Subjects who are likely to start taking drugs/medication on a chronic basis or that will undergo surgery during the trial.
* Subjects engaged in donation or who were recipients of blood products within 90 days before the start of the study.
* Subjects with alcohol use of more than 2 alcoholic beverages per day within the past month.
* Subjects participated in a clinical trial with a medicinal, supplemental, nutraceutical or drug within the past two months prior to the first dose in the current study.
* Use of lipid, cholesterol and/or blood-sugar lowering agents (e.g. statins, fibrates, bile acid sequestrants, PCSK9 inhibitors, prescription-based nicotinic acid derivatives (e.g. niacin extended release), metformin, sulfonylureas, including fish oil). If participants take fish oil supplements, they will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects using anti-inflammatory drugs on a chronic basis (e.g. aspirin, ibuprofen, diclofenac, celecoxib, etc).
* Subjects using supplements or substances present in formulation (malate, fisetin, glucosamine, alpha ketoglutaric acid, glycine, theanine, Rhodiola rosea, hyaluronic acid, ginger extract, pterostilbene, lithium). Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects using supplements or substances similar as those used in the formulation (e.g. resveratrol (similar to pterostilbene) or quercetin (similar to fisetin)). Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects taking NAD boosters, like NMN, nicotinamide riboside (NR), high-dose niacin (nicotinic acid), high-dose vitamin B3, high-dose nicotinamide (niacinamide) within 21 days before the start of the trial. Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects taking supplements or drugs or nutraceuticals to improve skin, such as hyaluronic acid, collagen, chondroitin, glucosamine. Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects with clinically significant abnormal laboratory results at screening.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Appearance of Fine Lines and Wrinkles | 6 months
  Fine lines and wrinkles measured by high resolution photography (BTBP Clarity Pro) to measure wrinkle severity (combines depth and width). Measured by computer calculation.

SECONDARY OUTCOMES:
Appearance of facial redness | 6 months
  Change in the appearance of facial redness by high resolution photography (BTBP Clarity Pro) and measures intensity of facial redness. Measured by computer calculation
Appearance of facial pigmentation | 6 months
  Change in the appearance of facial pigmentation by high resolution photography (BTBP Clarity Pro) and measures intensity of facial pigmentation. Measured by computer calculation
Appearance of facial texture | 6 months
  Change in the appearance of facial texture by high resolution photography (BTBP Clarity Pro) and measures evenness of skin surface. Measured by computer calculation
Skin hydration | 6 months
  Skin hydration measured by non-invasive device
Skin elasticity | 6 months
  Skin viscoelasticity measured by non-invasive device
Fasting lipids | 6 months
  Change in fasting lipids (LDL, HDL)
Hemoglobin A1c | 6 months
  Change in Hemoglobin A1c
Ultra-sensitive CRP | 6 months
  Change in ultra-sensitive CRP
Blood pressure | 6 months
  Change in blood pressure (diastolic and systolic)
Mental health survey | 6 months
  Assessment of mental health status by survey
Subjective skin health survey | 6 months
  Subjective assessment of skin health by survey
Epigenetic signals | 6 months
  Evaluation of epigenetic expression changes

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States